CLINICAL TRIAL: NCT03254511
Title: The Effect of Addition of Enoxaparin to Neoadjuvant Chemoradiation of Esophageal Cancer on the Clinical and Pathologic Response
Brief Title: Addition of Enoxaparin to Neoadjuvant Chemoradiation of Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyed Alireza Javadinia, Principal Investigator, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 941703; IRCT2016070628814N1 (Registry Identifier: the Iranian Registry of Clinical Trials)
Record Dates: First submitted 2017-08-11; First posted 2017-08-18 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Neoplasms
Keywords: neoadjuvant chemoradiation; pathologic response; low molecular weight heparin
MeSH Terms: conditions — Esophageal Neoplasms | interventions — enoxaparin sodium; Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enoxaparin (Experimental): In the enoxaparin group, patients are going to receive radiotherapy (median treatment dose will be 50.40 Gy in 25 to 32 fractions) with weekly concurrent chemotherapeutic combinations (paclitaxel [50 mg/m2] plus carboplatin [area under the carve=2]) with Enoxaparin Sodium 40 MG/0.2 ML Subcutaneous Injectable (40 mg daily).
  Interventions: Drug: Enoxaparin Sodium 40 MG/0.2 ML Subcutaneous Injectable; Radiation: Radiotherapy; Drug: Chemotherapeutic Combinations
- control (Active Comparator): In the control group, patients are going to receive radiotherapy (median treatment dose will be 50.40 Gy in 25 to 32 fractions) with weekly concurrent chemotherapeutic combinations (paclitaxel [50 mg/m2] plus carboplatin [area under the carve=2]) alone.
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapeutic Combinations

INTERVENTIONS:
Drug: Enoxaparin Sodium 40 MG/0.2 ML Subcutaneous Injectable — Patients are going to receive subcutaneouse Enoxaparin (40 mg daily).
  Arms: enoxaparin
Radiation: Radiotherapy — Patients will be treated with 3D conformal radiotherapy. The median treatment dose will be 50.40 Gy in 25 to 32 fractions.
Drug: Chemotherapeutic Combinations — Patients are going to receive weekly chemotherapy (paclitaxel [50 mg/m2] plus carboplatin [area under the carve=2]).

SUMMARY:
This is a randomized, single blind, multi-center, phase two clinical trial. Inclusion criteria are consist of non-metastatic esophageal cancer who are going to receive chemo-radiotherapy. Sample size is 100 people (50 people in each group). In the intervention group, patients are going to inject an enoxaparin (40 mg) daily concurrent by chemo-radiation. Therefore patients with esophageal cancer are going to assign randomly to control group (only chemo-radiotherapy) and intervention group (chemo-radiotherapy+enoxaparin) using 1:1 allocation. Four to 6 weeks after treatment, all patients undergo upper GI endoscopy and then esophagectomy. Endoscopic and pathological findings (after esophagectomy) are considered as clinical and pathological response, respectively.

DETAILED DESCRIPTION:
This is a randomized, single blind, multi-center, phase two clinical trial. Inclusion criteria are consist of non-metastatic esophageal cancer who are going to receive chemo-radiotherapy. One hundred patients are going to assign randomly by blocked randomized allocation (1:1) to receive radiotherapy (median treatment dose will be 50.40 Gy in 25 to 32 fractions) with weekly concurrent chemotherapy (paclitaxel [50 mg/m2] plus carboplatin [area under the carve=2]) with or without enoxaparin (40 mg daily). During radiotherapy and before each course of chemotherapy, all patients are going to visit by physician and complete blood count will be checked. All patients are going to undergo gastrointestinal endoscopy and then esophagectomy, 4-6 months after completion of chemo-radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnoses of esophageal squamous cell carcinoma by pathological evaluation
* Non-metastatic esophageal cancer
* Patient who are candidate for chemo-radiation treatment
* Normal complete blood count
* Normal kidney function test
* Normal liver function test
* Normal fasting blood sugar

Exclusion Criteria:

* Previous history of chest wall radiotherapy
* Previous history of chemotherapy
* Past medical history of Hypertension, diabetes mellitus, renal failure and liver failure
* Pathological report of adenocarcinoma or small cell carcinoma, neoplasm of other organs
* Discontent for the study
* Inability to do daily radiotherapy
* Unwillingness to esophagectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07-22 (Actual); Primary Completion 2017-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
clinical response | up to 6 weeks
  according to endoscopic findings (no lesion, primary lesion or became smaller less than 50%of primary lesion, become smaller more than 50% of primary lesion)
pathologic response | up to 6 weeks
  according to pathologic findings of esophageus specimen (complete Vs incomplete)
R staging (residual of tumor) | up to 6 weeks
  according to surgeon findings when esophagectomy is done (gross residue, microscopic residue, without residue)

SECONDARY OUTCOMES:
heparin induced thrombocytopenia | through study completion, an average of 5 weeks
  according to complete blood count

CONTACTS AND LOCATIONS:
Overall Officials: Ali Taghizadeh Kermani, M.D., Study Chair — Omid Hospital, Mashhad University of Medical Sciences, Mashhad, Iran; Sareh Hosseini, M.D., Study Director — Omid Hospital, Mashhad University of Medical Sciences, Mashhad, Iran; Seyed Alireza Javadinia, M.D., Principal Investigator — Omid Hospital, Mashhad University of Medical Sciences, Mashhad, Iran; Arezoo Gholami, M.D., Principal Investigator — Omid Hospital, Mashhad University of Medical Sciences, Mashhad, Iran
Locations (1):
- Mashhad University of Medical Sciences, Mashhad, Khorasan Razavi, Iran

IPD SHARING:
Plan to Share IPD: Undecided